CLINICAL TRIAL: NCT02315508
Title: A Balanced Randomised Placebo Controlled Double-blind Phase IIa Study to Investigate the Efficacy and Safety of AUT00063 Versus Placebo in Subjective Tinnitus
Brief Title: Evaluating Possible Improvement in Tinnitus Severity After 28 Days Dosing of the Study Drug AUT00063 Compared to Placebo
Acronym: QUIET-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUT032063
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — AUT00063

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AUT00063 (Experimental): 4 capsules of 200 mg of the new medicine, AUT00063, to take orally with food for 4 weeks.
  Interventions: Drug: AUT00063
- Placebo (Placebo Comparator): 4 capsules of placebo, to take orally with food for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUT00063 — 800 mg orally, once a day, for 4 weeks
  Other Names: Experimental
  Arms: AUT00063
Drug: Placebo — orally, once a day, for 4 weeks
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
This study aims to demonstrate that the new medicine AUT00063 is effective and safe in the treatment of tinnitus.

DETAILED DESCRIPTION:
Reduced activity at certain sites in the brain (called "voltage-gated potassium channels") has been linked to hearing problems, like age-related loss of hearing or tinnitus (a 'ringing' or buzzing noise in the ears).

AUT00063 is an experimental new medicine that has been developed to improve the action of these specific channels and so treat the brain component of these hearing problems.

The main purpose of this study is to try to demonstrate an improvement in the severity of tinnitus after 4 weeks of treatment with the study medicine or the placebo (dummy drug which does not contain the medication). Subjects will undergo a safety follow-up after the treatment period.

Safety and efficacy will be determined by looking at a number of assessments (physical examinations, blood sampling, hearing assessments, questionnaires, etc.) and in case of any serious medical event during the study. The amount of drug in the blood will also be measured.

It is expected that up to 152 people with tinnitus may take part in the study. The study participants will be recruited at around 16 Hospital sites in the UK.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking, who are UK residents registered with a UK General Practitioner;
* Experiencing stable tinnitus (consistent from day to day)
* Tinnitus has existed for not less than 6 months, and not more than 18 months - Contraceptive methods must be used before and for at least 30 days after the stop of the study treatment.

Exclusion Criteria:

* Severe hearing impairment such that verbal communication is unreliable;
* History of important cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases deemed clinically significant at the time of the study by the Investigator and which might be jeopardised by entering the study;
* Moderate or severe depression or generalised anxiety
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days of starting the investigational treatment
* Participation in hearing study, involving an intervention, within 3 months from last study visit;
* Central nervous system pathologies e.g. Multiple Sclerosis, Parkinson's disease;
* Tinnitus as a concomitant symptom of a known otological condition (including but not limited to otitis externa, otitis media, otosclerosis, cholesteatoma, Ménière's disease or other vestibular problems, acoustic neuroma, or temporo-mandibular joint disorder);
* Pulsatile tinnitus (rhythmical sounds that often beat in time with the heartbeat);
* Intermittent tinnitus (comes and goes from one day to the next);
* Surgery or medical condition that might would be expected to significantly affect absorption of medicines;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in subjective Tinnitus after 4 weeks treatment | 28 days
  To compare the change from baseline (D1 to D28) of the Tinnitus Functional Index overall score between AUT00063 (800 mg) and placebo.

SECONDARY OUTCOMES:
To further investigate the safety and tolerability profile of repeat administration of AUT00063 (assessing vital signs, physical examination, laboratory exams and ECG) | 42 days
  To investigate the safety and tolerability of AUT00063 by assessing vital signs, physical examination, laboratory exams and ECG
Change in Tinnitus Loudness matching after 4 weeks of treatment | 28 days
  Changes from baseline (D1) at Day 28 between treatment groups in Tinnitus loudness matching (LM).
Pharmacokinetic of AUT00063 (Exposure of AUT00063 ng/ml, measured as AUT00063 plasma levels) | at day 28
  Exposure of AUT00063 ng/ml, measured as AUT00063 plasma levels at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jaydip Ray, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Birmingham University Hospital, Birmingham
  - Bradford Teaching Hospital, Bradford
  - Bristol Royal Infirmary, Bristol
  - Cambridge University Hospitals NHS Trust, Cambridge
  - Frimley Health NHS Foundation Trust, Frimley
  - University College London Hospital NHS Foundation Trust, London
  - The Pennine Acute Hospitals NHS Trust, Manchester
  - Freeman Hospital, Newcastle
  - Norfolk and Norwich University Hospital Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Plymouth NHS Trust, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Salford Royal Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield, Sheffield
  - Lister Hospital, Stevenage
  - University Hospital of North Staffordshire, Stoke-on-Trent
  - Shrewsbury and Telford Hospital NHS Trust, Telford
  - Wrightington Hospital, Wigan

REFERENCES:
- [Derived] Hall DA, Ray J, Watson J, Sharman A, Hutchison J, Harris P, Daniel M, Millar B, Large CH. A balanced randomised placebo controlled blinded phase IIa multi-centre study to investigate the efficacy and safety of AUT00063 versus placebo in subjective tinnitus: The QUIET-1 trial. Hear Res. 2019 Jun;377:153-166. doi: 10.1016/j.heares.2019.03.018. Epub 2019 Mar 27. PMID 30939361